CLINICAL TRIAL: NCT01246726
Title: The Tumour Bed as Target for Breast Irradiation Following Breast Conserving Surgery
Brief Title: Multiple Oncological Serial Scans Study
Acronym: MOSS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: MRI scanner de-commissioned and there was no suitable alternative.
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: Bosum Buddies (Unknown); Friends of the Bristol Haematology and Oncology Centre (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ON/2009/3235
Record Dates: First submitted 2010-03-31; First posted 2010-11-23 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
Keywords: cancer, breast, radiotherapy, boost
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: CT SCAN — Prior to radiotherapy + after radiotherapy completion
Procedure: MRI scan — Prior to radiotherapy + after completion of radiotherapy
Procedure: 3D Ultrasound scan — Prior to radiotherapy + after completion of radiotherapy

SUMMARY:
This is a pilot study comparing the appearance and volume of the post surgical region in the intact breast, as determined by 3 modalities: computed Xray tomography (CT), 3 Dimensional ultrasound (USS), Magnetic resonance imaging (MRI) after breast conserving surgery and during whole breast irradiation.

DETAILED DESCRIPTION:
Consenting patients who have undergone breast conserving surgery and who are planned to receive radiotherapy will have their first MRI and CT scan within 2 weeks of treatment planning. This will be followed by 3 weeks radiotherapy treatment. 3D ultrasound scans will be performed in the first 2 weeks before radiotherapy, during the 2nd and 3rd weeks of radiotherapy and in the 2 weeks following radiotherapy.Following the radiotherapy patients will undergo both CT and MRI scans within 2 weeks of treatment completion.The whole process should take approximately 10 weeks.In this study the CT scans, MRI scan + USS are above standard care and are the additional interventions in this study group.

ELIGIBILITY:
Inclusion Criteria:

All female patients who, after breast conserving surgery, are to undergo whole breast irradiation with or without a boost. Ten patients will be for planned radiotherapy following both breast conservation surgery and chemotherapy and ten will be for planned radiotherapy following breast conservation surgery alone aged between 18 and 80years.

-

Exclusion Criteria:

Mastectomy T3 or T4 and N3 cases Patients who have not undergone surgery Severely claustrophobic patients Patients unable to lie flat Patients with any contraindications to MRI

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Maximal dimensions of post operative complex will be obtained using the British Colombia Cancer Agency Seroma Clarity score scale. | Within 3 months of radiotherapy completion
  Each modality of investigation i.e. CT, MRI +USS will be evaluated using the Seroma clarity score scale to determine the most useful investigational tool.

CONTACTS AND LOCATIONS:
Overall Officials: Amit K Bahl, MD,MRCP,FRCR, Principal Investigator — University Hospitals Bristol and Weston NHS Foundation Trust
Locations (1):
- University Hospitals Bristol NHS Foundation trust, Bristol, Bristol, United Kingdom